CLINICAL TRIAL: NCT00454285
Title: Bacteremia From Dental Extractions vs. Oral Hygiene
Brief Title: Bacteria Entering the Blood Stream From Tooth Extractions and Tooth Brushing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13559; R01DE013559-01 (NIH); 1R01DE013559-01A2 (NIH)
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2009-12

CONDITIONS: Bacteremia
Keywords: bacteremia,cultures, infective endocarditis, prophylaxis
MeSH Terms: conditions — Bacteremia; Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Effect of Amoxicillin on bacteremia following a single-tooth extraction — Administer Amoxicillin 1 hour prior to single-tooth extraction.

SUMMARY:
The major purposes of this prospective, randomized, clinical study are to:

1. Determine and compare the true incidence, nature, magnitude, and duration (INMD) of bacteremia (bacteria found in the bloodstream) resulting from a highly invasive dental office procedure (tooth extraction) and a minimally invasive and naturally occurring source of bacteremia (tooth brushing);
2. Measure the effect of the American Heart Association's guidelines for amoxicillin prophylaxis (preventive treatment) on the INMD of bacteremia resulting from a single tooth extraction.

DETAILED DESCRIPTION:
The use of antibiotic prophylaxis to prevent distant site infections (DSI) from oral pathogens remains a controversial issue in clinical practice. Little is known about the incidence, nature, and duration (IND) of bacteremia resulting from dental extractions or tooth brushing, either in the presence or absence of prophylactic antibiotic coverage. The purpose of this prospective, randomized, clinical study of 300 subjects is to characterize the bacteremia resulting from a highly invasive (single extraction) dental office procedure and a minimally invasive and naturally occurring source of bacteremia (i.e., tooth brushing). Subjects will be randomized into three equal groups: extraction with amoxicillin, extraction with placebo, and oral hygiene. The major goals are to: 1) improve our understanding of the IND of bacteremias from 10 specific oral pathogens (S. mitis, S. sanguis, S. oralis, S. intermedius, S. mutans, S. salivarius, F. nucleatum, A. Actinomycetemcomitans, E. corrodens and P. gingivalis) that have been reported to cause DSI; 2) measure the effect of the American Heart Association's guidelines for amoxicillin prophylaxis on the IND of bacteremia resulting from a single dental extraction. Blood for aerobic and anaerobic cultures will be drawn at six time points before, during, and following these oral procedures. We will employ a highly sensitive broth-based culturing system (i.e., BACTEC) and improve the specificity of the BACTEC results with the use of PCR sequence analysis. Detailed clinical information on the extent of disease in and around the involved teeth will determine the significance of local disease factors on the IND of the bacteremia from oral pathogens. Data from this study should have implications regarding future guidelines and standards of care concerning antibiotic prophylaxis for individuals currently felt to be at risk for DSI.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have at least 10 teeth and the need for a dental extraction.
* Subjects will be accepted into the study regardless of the extent of their odontogenic and/or periodontal disease, to include Type I through IV American Association of Periodontists classification.

Exclusion criteria:

* Subjects who need surgical extractions that require initial removal of bone overlying the surface of a tooth.
* Subjects who have taken systemic antibiotics within the previous 2 weeks.
* Subjects who require antibiotic coverage, based on current practice guidelines, prior to invasive dental procedures (e.g., cardiac valve abnormalities).

.Subjects with active viral infectious disease (e.g., hepatitis).

* Subjects who are immunocompromised (e.g., organ transplant, HIV).
* Subjects classified as American Society of Anesthesiology Class III or higher (i.e., a patient with poorly-controlled systemic disease).
* Subjects with facial cellulitis.
* Subjects who have had any manipulation of the gingiva within 1 hr prior to the study(e.g., eating, tooth brushing, chewing gum).
* Subjects with a history of penicillin allergy.
* Subjects deemed by the clinician to have a bacterial infection.
* Subjects with a temperature of 100.5 degrees Fahrenheit or above.
* Venous access unavailable in non-dominant arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2003-01; Primary Completion 2005-11 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall incidence of bacteremia in three groups | Blood Draws at 0, 2.5, and 5 minutes; and at 20. 40, and 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B. Lockhart,, DDS, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center Dental Clinic, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Lockhart PB, Brennan MT, Thornhill M, Michalowicz BS, Noll J, Bahrani-Mougeot FK, Sasser HC. Poor oral hygiene as a risk factor for infective endocarditis-related bacteremia. J Am Dent Assoc. 2009 Oct;140(10):1238-44. doi: 10.14219/jada.archive.2009.0046. PMID 19797553